CLINICAL TRIAL: NCT05970887
Title: Immunogenicity and Safety of Concomitant Administration of Omicron-containing Bivalent COVID-19 Vaccines With Seasonal Influenza Vaccines
Brief Title: Immunogenicity and Safety of Concomitant Administration of Bivalent COVID-19 Vaccines With Influenza Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic Kwandong University (Other)
Collaborators: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Min Joo Choi, Assistant Professor, Catholic Kwandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IS22OISE0060
Record Dates: First submitted 2023-07-28; First posted 2023-08-01 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Immune Response; Safety
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized clinical cohort study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- C group (Experimental): Concomitant administration of bivalent mRNA COVID-19 booster and quadrivalent influenza vaccination
  Interventions: Biological: bivalent BNT162b2 mRNA original/omicron BA.4-5 vaccine; Biological: quadrivalent influenza vaccine
- S group (COVID-19 vaccine only) (Placebo Comparator): separate administration of influenza vaccination followed by bivalent BA.4/BA.5 mRNA booster ≥4 weeks later
  Interventions: Biological: bivalent BNT162b2 mRNA original/omicron BA.4-5 vaccine
- S group (influenza vaccine only) (Placebo Comparator): separate administration of influenza vaccination followed by bivalent BA.4/BA.5 mRNA booster ≥4 weeks later
  Interventions: Biological: quadrivalent influenza vaccine

INTERVENTIONS:
Biological: bivalent BNT162b2 mRNA original/omicron BA.4-5 vaccine — The bivalent BNT162b2 mRNA original/omicron BA.4-5 vaccine is a combination of 15-µg of mRNA encoding the wild-type (WT) spike protein and 15-µg of mRNA encoding the spike protein of the Omicron BA.4/BA.5 subvariant.
  Arms: C group; S group (COVID-19 vaccine only)
Biological: quadrivalent influenza vaccine — The quadrivalent influenza vaccine is an inactivated vaccine containing 15μg HA/strain in each 0.5-mL dose, containing four influenza vaccine strains from the 2022-2023 northern hemisphere season
  Arms: C group; S group (influenza vaccine only)

SUMMARY:
The goal is to evaluate the immunogenicity and safety of coadministration of a bivalent BA.4/BA.5-adapted COVID-19 booster vaccine, and influenza vaccine among healthy adults during 2022-23 season.

DETAILED DESCRIPTION:
This was an open-label, non-randomized clinical trial conducted at the International St. Mary's Hospital in Incheon, South Korea. This study included two study groups: Concomitant administration of bivalent BA.4/BA.5 mRNA COVID-19 booster and quadrivalent influenza vaccination (QIV) and separate administration of influenza vaccination followed by bivalent BA.4/BA.5 mRNA booster ≥4 weeks later

* immunogenicity analysis : Blood was drawn at baseline and follow-up visit 4 weeks (day 28±7) after immunization.
* safety analysis : At 7 days after each vaccine dose, the participants were requested to record the occurrence, severity of solicited adverse events (AEs) through a standardized electronic questionnaire. Participants were also asked to record any unsolicited AEs during the 28 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* who agreed to receive both bivalent booster COVID-19 vaccine and influenza vaccine
* Only individuals who had passed at least 3 months after the last confirmation of SARS-CoV-2 infection and/or the third dose of COVID-19 vaccination

Exclusion Criteria:

* Individuals with a contraindication to any of the vaccine compounds were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
seroconversion rate of anti-severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike (S) immunoglobulin (IgG) between the C and S groups | at 28 days after booster dose
  seroconversion rate of anti-SARS-CoV-2 S IgG

SECONDARY OUTCOMES:
seroconversion rate of neutralizing antibody against SARS-CoV-2 | at 28 days after booster dose
  seroconversion rate of neutralizing antibody against wild type, Omicron BA.5
geometric mean titer against SARS-CoV-2 | at 28 days after booster dose
  geometric mean titer against SARS-CoV-2 (Anti-S IgG, neutralizing antibody)
seroconversion rate of four influenza strains | at 28 days after immunization
  seroconversion rate of four influenza strains
seropositive rate of four influenza strains | at 28 days after immunization
  seropositive rate of four influenza strains
geometric mean titer against four influenza strain | at 28 days after immunization
  geometric mean titer against four influenza strain
The incidence rate of adverse events (AEs) | within 28 days
  The incidence rate of AEs within 7 days, AEs within 28 days, and serious AEs

CONTACTS AND LOCATIONS:
Overall Officials: Min Joo Choi, Doctor, Principal Investigator — International St. Mary's Hospital
Locations (1):
- International St. Mary's hospital, Incheon, Seo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No